CLINICAL TRIAL: NCT03870178
Title: Effects of tDCS on Maximal Isometric Strength and Endurance Test of Trunk Extensors in Healthy Subjects.
Brief Title: Effects of tDCS on Maximal Isometric Strength and Endurance Test of Trunk Extensors.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade Federal do Piauí (Other)
Responsible Party: Principal Investigator, Fuad Ahmad Hazime, Clinical Professor - Physical Therapy Department, Universidade Federal do Piauí
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1.577.037
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Healthy
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Active Comparator): Anodal tDCS over trunk motor cortex representation. Intensity: 2mA Time: 20 minutes
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Sham tDCS (Sham Comparator): Anodal tDCS over trunk motor cortex representation. Itensity: 2mA Time: 20 minutes (30s ON)
  Interventions: Device: Transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — The noninvasive and nonpharmacological weak electrical current applied to the scalp to modulate cortical excitability.

SUMMARY:
Improving trunk muscle strength and endurance is one of the many goals to be achieved in rehabilitation protocols for a variety of health conditions. Cerebral electrical stimulations techniques, such as transcranial direct current stimulation (tDCS) can modulate motor brain areas involved in motor functions. However, their effects on trunk function are lacking.

This study aims to investigate the effects of transcranial direct current stimulation (tDCS) on trunk muscle strength and endurance in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with no complaints of pain, discomfort in the musculoskeletal system.

Exclusion Criteria:

* Musculoskeletal or neurological disorder
* Under medication

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Isometric trunk extension | Pre and Post-test (immediately after tDCS)
  Maximal isometric voluntary contraction (Kgf)
Trunk muscle endurance | Pre and Post-test (immediately after tDCS)
  Time to task failure (TTF) on the Sorensen test

SECONDARY OUTCOMES:
Isometric trunk extension | 15 minutes post-stimulation
  Maximal isometric voluntary contraction (Kgf)
Isometric trunk extension | 30 minutes post-stimulation
  Maximal isometric voluntary contraction (Kgf)
Trunk muscle endurance | 15 minutes post-stimulation
  Time to task failure (TTF) on the Sorensen test
Trunk muscle endurance | 30 minutes post-stimulation
  Time to task failure (TTF) on the Sorensen test

CONTACTS AND LOCATIONS:
Overall Officials: Fuad Hazime, PhD, Principal Investigator — Department of Physical Therapy. Federal University of Piaui
Locations (1):
- Department of Physical Therapy. Federal University of Piaui, Parnaíba, Piauí, Brazil